CLINICAL TRIAL: NCT01681199
Title: The Efficacy of Lescol XL(Fluvastatin Extended Release 80 mg) on Atherosclerosis Progression in Patients With Newly Diagnosed Coronary Heart Disease
Brief Title: Fluvastatin AmelIorates aTHerosclerosis Study
Acronym: FAITH
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Chang sheng Ma, director of cardiology department, Beijing Anzhen Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AZYY-XNK-2012001
Record Dates: First submitted 2012-09-05; First posted 2012-09-07 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Coronary Heart Disease; Atherosclerosis
Keywords: statin; atherosclerosis; Coronary heart disease; OPN; OPG
MeSH Terms: conditions — Coronary Disease; Atherosclerosis | interventions — Fluvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fluvastatin extended release tablet (Experimental): Fluvastatin extended release tablet 80mg/day
  Interventions: Drug: Fluvastatin extended release tablet

INTERVENTIONS:
Drug: Fluvastatin extended release tablet
  Other Names: Lescol XL

SUMMARY:
The study is designed to assess the effect of statin on atherosclesrosis progression as well as to explore its potential mechanism besides lipid modifying , such as effect on inflammation and vascular calcification.

DETAILED DESCRIPTION:
Carotid IMT has been used in various studies (e.g. ASAP, ARBITER, METEOR) and is well accepted as a valid surrogate marker for atherosclerosis. The thickness of CIMT is significantly associated with the presence and the extent of coronary disease. Slower progression of atherosclerosis as measured by carotid ultrasound is also associated with a lower risk of nonfatal MI. In a meta analysis, for every 0.0 1-mm-per-year decrease in carotid IMT, there was a significant 18% reduction in the risk of nonfatal MI. Measurement of carotid IMT carries the advantage of being non-invasive and easy to use with a good degree of reproducibility.

Statins have been shown to slow the progression of atherosclerosis or even to induce regression of atherosclerosis. Change of carotid IMT by statins have been found to correlate with the extent of LDL-C reduction and HDL-C increase however non-lipid effects (e.g. effects on inflammation, calcification ) may also play a role in the beneficial effects of statins on atherosclerosis.Osteopontin (OPN), an acidic phosphoprotein, and osteoprotegerin (OPG), a member of the tumor necrosis factor-a receptor superfamily, have been recently demonstrated to modulate vascular calcification. Recent studies have shown an association of serum OPN and OPG levels with cardiovascular diseases and vulnerable carotid plaque .

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed coronary heart disease
2. One or more maximum IMT measurements of ≥1.1mm.
3. Age 45 to 70 years old
4. LDL-C≥130mg/dL
5. Not receiving regular lipid lowering treatment
6. Written Informed Consent

Exclusion Criteria:

1. Myocardial infarction as the first symptoms of coronary heart disease
2. Patients with known hypersensitivity to fluvastatin or any of the excipients
3. Pregnancy or lactation, or women of childbearing potential not using effective contraception
4. Known muscle disease or history of muscle disease (e.g. myopathy, myositis, rhabdomyolysis) and/or serum CK levels greater than 2 x upper limit of normal (ULN)
5. renal dysfunction
6. Active liver disease and/or serum transaminase levels (ALT, AST) greater than 2x ULN
7. Any conditions the investigator consider not suitable for long-term follow up

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-04 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
carotid IMT | 1 year

SECONDARY OUTCOMES:
lipid variables:TC, TG, LDL-C, HDL-C, apo B, apo A-I | week 12 and 24

OTHER OUTCOMES:
hs-CRP, Lp-PLA2, OPN and OPG. | week 12,24 and 52

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiology department ,Beijing Anzhen hospital, Beijing, Beijing Municipality, China